CLINICAL TRIAL: NCT06869447
Title: Lung Cancer Better Breathing Study
Brief Title: New York Better Breathing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: I-3969424; NCI-2025-01035 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3969424 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Localized Lung Carcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patients will be blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (moderate/high intensity RMT) (Experimental): Patients participate in home-based/virtually supervised and unsupervised moderate/high intensity RMT sessions consisting of three sets of 15 breaths using the Power Lung device over 20 to 30 minutes per session, 5 days per week for 12 weeks. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Procedure: Respiratory Muscle Training
- Group II (low intensity sham RMT) (Sham Comparator): Patients participate in home-based/virtually supervised and unsupervised low intensity sham RMT sessions using the Power Lung breathing device over 20 to 30 minutes per session, 5 days per week for 12 weeks. Patients also undergo blood sample collection throughout the study. Patients may optionally participate in the moderate/high intensity RMT session for 6 weeks upon study completion.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Procedure: Sham Intervention

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Other: Medical Device Usage and Evaluation — Use Power Lung breathing device
Other: Questionnaire Administration — Ancillary studies
Procedure: Respiratory Muscle Training — Participate in RMT sessions
  Other Names: RMT
  Arms: Group I (moderate/high intensity RMT)
Procedure: Sham Intervention — Participate in sham sessions
  Other Names: Sham Comparator
  Arms: Group II (low intensity sham RMT)

SUMMARY:
This clinical trial evaluates the effects of whether breathing exercises at home can reduce symptoms and help stage I-III lung cancer survivors stay active. Over 70% of lung cancer survivors have trouble breathing, feel tired, and have lower levels of fitness. This is often because their breathing muscles are weaker after surgery. Many survivors find it hard to exercise, which affects their quality of life and overall survival. A training program to strengthen these muscles might reduce breathing problems, lower fatigue, and improve quality of life. Staying active could also help boost the immune system to fight cancer. Respiratory muscle training (RMT) involves a series of breathing and other exercises that are performed to improve the function of the respiratory muscles through resistance and endurance training. Participating in a home-based RMT intervention may reduce symptoms from cancer or treatment in lung cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of delivering a home-based RMT program to Black and White lung cancer survivors.

II. Determine the effects of RMT on symptom management (quality of life [QoL], fatigue, dyspnea, sleep, etc.), performance (respiratory muscle and lower extremity strength), and physical activity in Black and White lung cancer survivors.

III. Determine if RMT improves cancer related anti-tumor activity (T-cell function) and diminishes markers of immunosuppression (myeloid-derived suppressor cells [MDSCs], regulatory T cells) and inflammation (high-sensitivity C-reactive protein, (hsCRP) in circulation.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients participate in home-based/virtually supervised and unsupervised moderate/high intensity RMT sessions consisting of three sets of 15 breaths using the Power Lung device over 20 to 30 minutes per session, 5 days per week for 12 weeks. Patients also undergo blood sample collection throughout the study.

GROUP II: Patients participate in home-based/virtually supervised and unsupervised low intensity sham RMT sessions using the Power Lung breathing device over 20 to 30 minutes per session, 5 days per week for 12 weeks. Patients also undergo blood sample collection throughout the study. Patients may optionally participate in the moderate/high intensity RMT session for 6 weeks upon study completion.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Able to speak, read and comprehend the English language
* Self-identify as non-Hispanic Black or White.
* Are < 15 months of histologically confirmed invasive, non-metastatic, lung cancer diagnosis.
* Have received surgical treatment (primarily stage I, II and III) and have completed all cancer treatments (surgery, chemotherapy, radiation).
* Willing to provide biospecimen samples for the study (blood) which will be collected in the comfort of the patient's home by a mobile phlebotomy group.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Participant is metastatic (stage IV) at study entry.
* Has contraindications for respiratory muscle training (e.g., recent pulmonary embolism, aortic aneurysm, current pneumothorax).
* Is actively engaging in a structured exercise program and/or meeting exercise guidelines.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who complete at least 3 respiratory muscle training (RMT) sessions/week (Compliance) (Aim 1) | Up to 12 weeks
  Compliance will be estimated using 90% confidence intervals (CIs) obtained by Jeffreys' prior method. Will be modeled as a function of time (e.g., week) and prespecified exogenous factors (e.g., baseline age, pre-intervention dyspnea scores, self-reported history of exercise, lung cancer treatment received, treatment side-effects) using a GEE (Generalized Estimating Equations) logistic regression model (autoregressive covariance structure). Will also be explored with data stratified by race and gender.
Proportion of planned sessions completed (Adherence) (Aim 1) | Up to 12 weeks
  Adherence will be defined as the number of sessions completed divided by the total number of sessions planned (70% of the 42/60 sessions). Will be estimated using 90% CIs obtained by Jeffreys' prior method. Will also be explored with data stratified by race and gender.
Proportion of total completed to total planned cumulative dose (Tolerability) (Aim 1) | Up to 12 weeks
  Tolerability ratio will be assessed using Relative Dose Intensity and rate of lost to follow-up and discontinuation.
Inspiratory muscle strength (Aim 2) | Up to 12 weeks
  Will perform remote respiratory muscle strength testing with a handheld device (Leaton, China) to measure diaphragm strength. All will be done per American Thoracic Society guidelines. A minimum of 3 trials with 5% of each will be required. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using linear mixed models (LMMs).
Change in dyspnea (Aim 2)-Dyspnea-12 survey | Through study completion up to 7 months
  Will be measured using the Dyspnea-12 survey survey that measures recent breathlessness with 12 questions related to dyspnea, each evaluated on a scale of 0-4 (0=none, 1=mild, 2=moderate, 3=severe) that indicate how troubled people are by each of these 12 topics, for a total possible score ranging from 0 to 36, where lower scores relate to better outcomes.- Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in dyspena (Aim 2)- Functional Assessment of Chronic Illness Therapy (FACIT) dyspnea | Through study completion up to 7 months
  the Functional Assessment of Chronic Illness Therapy (FACIT) dyspnea questionnaire. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in cancer-related fatigue (Aim 2) - Brief Fatigue Inventory | Through study completion up to 7 months
  This 9-item scale assesses the severity and interference of fatigue based on a 0 (no fatigue) to 10 (greatest fatigue) scale
Change in cancer related Fatigue (Aim 2) - FACIT fatigue scale | Through study completion up to 7 months
  s a 13-item patient-reported measure of fatigue. Items are scored on a 0 - 4 response scale with anchors ranging from "Not at all" to "Very much so".
Circulating levels of myeloid-derived suppressor cells (MDSCs) (Aim 3) | Prior to start of 12 week program and after the end of the 12 week program
  All flow cytometry assessments will be performed in the Flow & Image Cytometry Shared Resource (FICSR). A key outcome will be the quantification of immunosuppressive MDSCs, which play an important role in lung cancer prognosis. Myeloid cells (CD45+ CD11b+CD33+) will be assessed for both major human MDSC subsets, polymorphonuclear myeloid-derived suppressor cells, and monocytic MDSCs. For analysis of peripheral blood mononuclear cells, cells will first be collected over a Ficoll-Hypaque gradient, where both MDSC subsets, as well as all other immune populations analyzed will reside. Polymorphonuclear-MDSCs will be defined as CD11b+CD33+HLA-DR-CD14-CD15+CD66b+, whereas M-MDSCs will be defined as CD11b+CD33+HLA-DRlo/- CD14+CD15-CD66b-.
Circulating levels conventional T cell populations (CD3+) (Aim 3) | Prior to start of 12 week program and after the end of the 12 week program
  All flow cytometry assessments will be performed in the FICSR. Will be stratified based on CD4 or CD8 expression, and will be further defined by their differentiation, activation, or exhaustion states.

SECONDARY OUTCOMES:
Proportion of eligible patients who elected to participate in the trial (Acceptability) (Aim 1) | Up to 12 weeks
  Enrollment rate will be summarized using frequencies and relative frequencies overall and by race and ethnicity.
Attrition rate (Feasibility) (Aim 1) | At 6 and 12 weeks
  An acceptable attrition rate will be defined as < 20%.
Patient-reported barriers to and facilitators of participation and sustained participation (Feasibility) (Aim 1) | At 6 and 12 weeks
Barriers to and facilitators (Aim 1) | At 6 and 12 weeks
  Identified as important for influencing exercise behavior among cancer survivors will be examined by gender and race, particularly those identified by lung cancer survivors, including social determinants of health. Will primarily use quantifiable Likert scales to rate the importance of each facilitator and barrier. Open-ended items will be included to collect factors not captured through closed survey questions.
Satisfaction with RMT and RMT-sham sessions (Aim 1) | At 6 and 12 weeks
  Will be evaluated by a survey assessment using patient-reported satisfaction with different intervention components using 0 to 10 Likert rating scales.
Exercise related dyspnea (Aim 2) | Up to 3 months follow-up
  Will be assessed immediately following performance tests with the 0-10 Borg scale. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in general quality of life (QoL) (Aim 2) | Through study completion up to 7 months
  Will be assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-30. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in disease-specific QoL (Aim 2) | Through study completion up to 7 months
  Will be assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in 2-minute step test (Aim 2) | Through study completion up to 7 months
  Will be Will be assessed to measure cardiorespiratory fitness that correlates with the 6-minute walk test. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in 30 second sit-to-stand test (Aim 2) | Through study completion up to 7 months
  Will be assessed to measure lower extremity strength. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in sleep (Aim 2) | Through study completion up to 7 months
  Will be assessed using the Pittsburgh Sleep Quality Index and Epworth daytime sleepiness scale. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in leisure-time physical activity (Aim 2) | Through study completion up to 7 months
  Will be assessed using the Godin Leisure-Time Exercise Questionnaire. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in physical activity and daily steps (Aim 2) | Through study completion up to 7 months
  Will be objectively monitored with an activity tracker. Fitness trackers will be synchronized during weekly follow-ups. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in pain (Aim 2) | Through study completion up to 7 months
  Will be assessed using pain questions taken from the Patient-Reported Outcomes Measurement Information System-29 questionnaire which assess pain intensity and interference. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
Change in peak inspiratory and expiratory muscle strength (Aim 2) | Through study completion up to 7 months
  Will be assessed using pa hand-held monometer. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies. Baseline demographic and clinical characteristics may be compared between study arms using the Mann-Whitney U and Fisher's exact tests, as appropriate. Will also be assessed using LMMs.
High-sensitivity C-reactive protein (Aim 3) | Prior to start of 12 week program and after the end of the 12 week program
  Will be measured with a Roche COBAS 8000 chemistry analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Ray, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States